CLINICAL TRIAL: NCT04290455
Title: The Efficacy of Microblephararoexfoliation in the Treatment of Anterior Blepharitis
Brief Title: Treatment of Anterior Blepharitis With Microblepharoexfoliation Procedure
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of recruitment during COVID
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Saba K. Al-Hashimi, MD, Assistant Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20-000084
Record Dates: First submitted 2020-02-21; First posted 2020-03-02 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Anterior Blepharitis
MeSH Terms: interventions — Granulex

STUDY DESIGN:
Intervention Model Description: A prospective, randomized, paired-eye trial.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigators who assess outcomes of anterior blepharitis will not know the arms that patients are in
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment arm (Experimental): using the microblepharoexfoliative procedure
  Interventions: Device: Microblepharoexfoliative procedure with BlephEx™; Procedure: Daily eyelid cleansing with eyelid wipes (Optase)
- control arm (Active Comparator): using eyelid wipe (Optase)
  Interventions: Procedure: Eyelid cleansing with eyelid wipes (Optase); Procedure: Daily eyelid cleansing with eyelid wipes (Optase)

INTERVENTIONS:
Device: Microblepharoexfoliative procedure with BlephEx™ — The device will be used to clean both upper and lower eyelid in the office visit.
  Arms: treatment arm
Procedure: Eyelid cleansing with eyelid wipes (Optase) — Eyelid cleansing will be done with eyelid wipes (Optase) by one clinician
  Arms: control arm
Procedure: Daily eyelid cleansing with eyelid wipes (Optase) — Patients in both arms will be instructed to do self-eyelid cleansing with eyelid wipes (Optase) daily at home for 21 days

SUMMARY:
Objective: To investigate the efficacy of microblepharoexfoliation by BlephEx™ as an adjunct to eyelid cleansing in the treatment of anterior blepharitis and to validate the grading score of lid contamination to describe the severity of anterior blepharitis. Design: A prospective, randomized, paired-eye trial. Methods: One of patients' eyes will be randomized into the microblepharoexfoliation group which will use the BlephExTM device during the in-house lid cleansing procedure. The other eye will be in the control group which will receive conventional lid cleansing. The parameters indicating the efficacy of the microblepharoexfoliation procedure including the symptom scoring system; the Standard Patient Evaluation of Eye Dryness Questionnaire (SPEED), lashes contamination, lid margin redness, number of preservative free artificial tears used per day, meibomian gland quality and expressibility will be recorded at the screening visit and 3-week follow-up visit. The patient will be instructed to do warm compression and lid cleansing at home once a day with Optase eyelid scrubs for 3 weeks on both eyes before follow-up.

DETAILED DESCRIPTION:
This study will be prospective, randomized, paired eye trial. Twenty patients with symptomatic anterior blepharitis with or without meibomian gland dysfunction who have a lash contamination score >1 and the Standard Patient Evaluation of Eye Dryness Questionnaire score (SPEED score) >= 1 will be included in the study. The criteria for grading of lashes contamination is defined as: 0= Clear lashes, 1=Slight contamination (involvement of lashes >0 but <25%), 2=Mild (>=25% but < 50%), 3=Moderate (>=50% but < 75%), and 4=Severe (>=75%). Patients will be recruited from the Dry Eye Clinic, Jules Stein Eye Institute, UCLA. The informed consent will be obtained from each patient. Patients who have been given a topical corticosteroid within 6 weeks before entering the study or need a topical corticosteroid or topical antibiotics as an adjunct to lid cleansing will be excluded from the study. Patients with concurrent conjunctivitis or keratopathy will also be excluded. Previous topical medications before patients enter the study such as anti-glaucoma medications and artificial tears will be continued.

One of the patients' eyes will be simply randomized into the interventional group in which the BlephExTM device(1) will be used to perform eyelid margin and lash cleansing. The other eye will be entered into the control group in which eyelid cleansing in a conventional way will be done using Optase wipes. In the screening visit, the Standardized Patient Evaluation of Eye Dryness (SPEED) questionnaire score and eyelid contamination will be assessed to recruit eligible patients. Before eyelid cleansing, images of the eyelid margin will be obtained by Oculus Keratograph 5M, Wetzlar, Germany and will be used to grade lashes contamination and lid margin redness by two independent observers. Parameters of interest of each eye will be evaluated separately. The primary outcomes are symptoms which will be scored using the Standard Patient Evaluation of Eye Dryness Questionnaire (SPEED)(2) and lashes contamination which will be graded as described above. Other outcomes of interest are lid margin redness, and the number of preservative free artificial tears used per day. The lid margin redness is graded as 0=Clear/white 1=Slight redness 2=Mild redness 3=Moderate redness 4=Severe redness. Patients will also be evaluated for concurrent meibomian gland dysfunction by evaluating meibum quality and expressibility of meibomian glands according to the International Workshop on Meibomian Gland dysfunction 2011(3). Meibum quality is assessed in each of eight glands of the central third of the lower lid on a scale of 0 to 3 for each gland: 0, clear; 1, cloudy; 2, cloudy with debris (granular); and 3, thick, like toothpaste (total score range, 0-24). Expressibility is assessed on a scale of 0 to 3 in five glands in the lower or upper lid, according to the number of glands expressible: 0, all glands; 1, three to four glands; 2, one to two glands; and 3, no glands. Patients who have minimally altered secretion grade ≥ 2-4 and expressibility ≥ 1 will be diagnosed with MGD. The images of eyelids will be taken again immediately after eyelid cleansing and eyelid contamination scores will be evaluated. The patient will then be instructed to perform lid cleansing at home once a day with eyelid cleansing wipes (Optase) for 21 days. The technique will be demonstrated to the patient in clinic. The follow-up visits will be at 21 days. At the follow-up visit, all of the data obtained in the screening visit will be repeated.

ELIGIBILITY:
Inclusion Criteria:

- anterior blepharitis with or without meibomian gland dysfunction who have a lash contamination score >1 and the Standard Patient Evaluation of Eye Dryness Questionnaire score (SPEED score) >= 1

Exclusion Criteria:

* Patients who have been given a topical corticosteroid within 6 weeks before entering the study or need a topical corticosteroid or topical antibiotics as an adjunct to lid cleansing will be excluded from the study.
* Patients with concurrent conjunctivitis or keratopathy will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-06-02 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Change from the baseline of the Standardized Patient Evaluation of Eye Dryness (SPEED) questionnaire score 21 days after treatment | Day 21 after treatment
Change from the baseline grading of lashes contamination 21 days after treatment | Day 21 after treatment
  The criteria for grading of lashes contamination is defined as severity of debris on lashes: 0= Clear lashes, 1=Slight contamination (involvement of lashes >0 but <25%), 2=Mild (>=25% but < 50%), 3=Moderate (>=50% but < 75%), and 4=Severe (>=75%).

SECONDARY OUTCOMES:
Lid margin redness | Baseline and Day 21 after treatment
  The lid margin redness is graded as 0=Clear/white 1=Slight redness 2=Mild redness 3=Moderate redness 4=Severe redness.
Frequency of preservative-free artificial tear eye drops used per day | Baseline and Day 21 after treatment
Degree of meibomian gland dysfunction | Baseline and Day 21 after treatment
  Assessment of meibum quality and expressibility of meibomian gland according to the International Workshop on Meibomian Gland dysfunction 2011(3). Meibum quality is assessed in each of eight glands of the central third of the lower lid on a scale of 0 to 3 for each gland: 0, clear; 1, cloudy; 2, cloudy with debris (granular); and 3, thick, like toothpaste (total score range, 0-24). Expressibility is assessed on a scale of 0 to 3 in five glands in the lower or upper lid, according to the number of glands expressible: 0, all glands; 1, three to four glands; 2, one to two glands; and 3, no glands. Patients who have minimally altered secretion grade ≥ 2-4 and expressibility ≥ 1 will be diagnosed with MGD.

CONTACTS AND LOCATIONS:
Locations (1):
- Stein Eye Institute, UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ngo W, Situ P, Keir N, Korb D, Blackie C, Simpson T. Psychometric properties and validation of the Standard Patient Evaluation of Eye Dryness questionnaire. Cornea. 2013 Sep;32(9):1204-10. doi: 10.1097/ICO.0b013e318294b0c0. PMID 23846405
- [Background] Nichols KK, Foulks GN, Bron AJ, Glasgow BJ, Dogru M, Tsubota K, Lemp MA, Sullivan DA. The international workshop on meibomian gland dysfunction: executive summary. Invest Ophthalmol Vis Sci. 2011 Mar 30;52(4):1922-9. doi: 10.1167/iovs.10-6997a. No abstract available. PMID 21450913